CLINICAL TRIAL: NCT07101939
Title: A Two-part, Phase 2a Randomized, Part Parallel-group, Double-blind Placebo-controlled Cross-over Multi-center Study to Evaluate the Effect of Two Dose Levels of (S)-Pindolol Benzoate (ACM-001.1) on Lean Body Mass in Obese Patients During (PROACT 1), and Post-semaglutide Therapy (PROACT 2)
Brief Title: A Study of the Effect of (S)-Pindolol Benzoate (ACM-001.1) on Lean Body Mass (LBM) in Obese Patents During (PROACT 1), and Post-semaglutide Therapy (PROACT 2)
Acronym: PROACT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Actimed Therapeutics Ltd (Industry)
Collaborators: SCIRENT Clinical Research and Science d.o.o. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACM-001-2024-01-CT
Record Dates: First submitted 2025-06-20; First posted 2025-08-03 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Muscle Loss
Keywords: semaglutide; s-pindolol; obesity; glp-1; glucagon-like peptide-1 receptor agonist; lean body mass
MeSH Terms: conditions — Obesity; Muscular Atrophy | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: A two-part, randomized, part parallel-group, double-blind placebo-controlled cross-over multi-center study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 semaglutide, low dose ACM-001.1 or sham injection/placebo during semaglutide therapy PROACT 1 (Active Comparator): Patients in Arm 1 will be randomized to a crossover design, to receive either semaglutide and low dose ACM-001.1 BID or a sham injection and placebo ACM-001.1 BID during Period 1. Following washout, in Period 2 patients within Arm 1 and Arm 2 will cross-over onto the opposing treatment.
  Interventions: Drug: (S)-pindolol benzoate; Drug: Semaglutide; Drug: Placebo to (S)-pindolol benzoate
- Arm 2 semaglutide, high dose ACM-001.1 or sham injection/placebo during semaglutide therapy PROACT 1 (Active Comparator): Patients in Arm 2 will be randomized to a crossover design, to receive either semaglutide and high dose ACM-001.1 BID (Group 2a) or a sham injection and placebo ACM-001.1 BID (Group 2b) during Period 1. Following washout, in Period 2 patients within Arm 1 and Arm 2 will cross-over onto the opposing treatment.
  Interventions: Drug: (S)-pindolol benzoate; Drug: Semaglutide; Drug: Placebo to (S)-pindolol benzoate
- Arm 3 ACM-001.1 low dose, high dose or placebo following semaglutide therapy PROACT 2 (Active Comparator): Patients randomized to Arm 3 will receive semaglutide and placebo ACM-001.1 BID during Period 1. Patients in Arm 3 will be further randomised into one of three treatment groups for Period 2:
  Group 3a will receive a sham injection and low dose ACM-001.1 BID Group 3b will receive a sham injection and high dose ACM-001.1 BID Group 3c will receive a sham injection and Placebo ACM-001.1 BID
  Interventions: Drug: (S)-pindolol benzoate; Drug: Semaglutide; Drug: Placebo to (S)-pindolol benzoate

INTERVENTIONS:
Drug: (S)-pindolol benzoate — (S)-pindolol benzoate (ACM-001.1) immediate release tablet containing (S)-pindolol benzoate administered BID.
  Other Names: ACM-001.1
Drug: Semaglutide — Semaglutide, solution for injection in pre-filled pen
Drug: Placebo to (S)-pindolol benzoate — Placebo to ACM-001.1 immediate release tablet administered BID

SUMMARY:
Semaglutide is approved for weight management (weight loss and weight maintenance) in adult obese patients. Drug treatments like semaglutide that result in weight-loss can also decrease muscle mass. The purpose of this study is to investigate the effect of ACM-001.1 (the study drug) on how much muscle is lost when a person takes it with semaglutide (PROACT 1) and how much muscle mass is gained when a person continues taking ACM-001.1 but stops taking semaglutide (PROACT 2).

DETAILED DESCRIPTION:
The study will compare the effects of ACM-001.1 (the study drug) when it is taken at the same time as semaglutide, and after semaglutide treatment has stopped. To allow the measurement of the effect of each treatment type, the study will involve the use of a placebo tablet and a 'sham' (fake) injection of semaglutide.

Various tests will be used to measure the effect of the study drug. These will include a DEXA scan (like an X-ray). The study will also include measurements of weight, tests on the heart, and tests of muscle function. Questionnaires relating to health and well-being will also be used. Blood samples will be taken and tested to check overall health.

The study takes place in two parts, each lasting 20 weeks. Between each 20-week period) there is a 4-week 'wash-out' period during which patients will not receive any treatment.

ACM-001.1 (or placebo) is a tablet for oral administration (by mouth). Two doses of ACM-001.1 are being tested in this study. The semaglutide or sham injection will be administered once every week.

The study is 'double-blind', neither the patient or the doctor will know if the patient is taking ACM-001.1 or placebo or which dose they receive.

The total study is expected to run for approximately 18 months.

ELIGIBILITY:
Key Inclusion Criteria:

Eligible for treatment with semaglutide.

Have a BMI of ≥30.0 kg/m².

Key Exclusion Criteria:

Type 2 diabetes mellitus who in the preceding 90 days have either:

* received a GLP-1RA (including semaglutide),
* had a hypoglycaemic event,
* lost >5 kg weight,
* had a HBA1C over 10.0%.

Any cardiovascular event within previous 6 months, uncontrolled hypertension, known congestive heart failure, or angina during the past year

Known severe chronic obstructive pulmonary disease (COPD)

Concomitant use of beta blockers and patients with contra indications to beta blockers

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-23 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
The change in lean body mass (LBM) in patients receiving one of two doses of ACM-001.1 whilst also receiving semaglutide. | 20 weeks
  In Arms 1 and 2: The change in lean body mass (LBM) grams/4 weeks over 20 weeks comparing 2 doses of ACM-001.1 with placebo. Body composition parameters will be measured using Dual Energy X-ray absorptiometry (DEXA) scan.
The change in lean body mass (LBM) grams/4 weeks over 20 weeks following semaglutide treatment. | 20 weeks
  In Arm 3: The change in lean body mass (LBM) grams/4 weeks over 20 weeks comparing 2 doses of ACM-001.1 with placebo. Body composition parameters will be measured using Dual Energy X-ray absorptiometry (DEXA) scan.

SECONDARY OUTCOMES:
Changes in fat mass during and following semaglutide treatment | 20 weeks
  In Arms 1 & 2: The change in fat mass (grams/4 weeks) over 20 weeks during semaglutide treatment comparing 2 doses of ACM-001.1 with placebo will be measured by DEXA scan.
  In Arm 3: The change in fat mass (grams/4 weeks) following semaglutide therapy comparing 2 doses of ACM-001.1 with placebo will be measured by DEXA scan.
Muscle Strength (Handgrip strength) during and following semaglutide treatment | 20 weeks
  In Arms 1 & 2: The change in Handgrip strength (kg/100g of arm lean mass) over 20 weeks comparing 2 doses of ACM-001.1 with placebo.
  In Arm 3: The change in Handgrip strength (kg/100g of arm lean mass) over 20 weeks comparing 2 doses of ACM-001.1 with placebo.

OTHER OUTCOMES:
An evaluation of changes in body weight during and following semaglutide treatment | 20 weeks
  In Arms 1 & 2: An evaluation of changes in body weight (kg/4 weeks) as the change from baseline (Period 1) over 20 weeks comparing 2 doses of ACM-001.1 with placebo.
  In Arm 3: An evaluation of changes in body weight (kg/4 weeks) as the change from baseline at the end of semaglutide therapy comparing 2 doses of ACM-001.1 with placebo.
Change in lean body mass (LBM) at the end of semaglutide therapy comparing 2 doses of ACM-001.1 with placebo | 20 weeks
  In Arm 3: The change in lean body mass (LBM) (g/4 weeks) after completing a period of 20 weeks of semaglutide therapy (plus placebo) comparing 2 doses of ACM-001.1 with placebo
Evaluation of hip:waist ratio during and following semaglutide treatment | 20 weeks
  In Arms 1 & 2: An evaluation of changes in hip:waist ratio (each circumference measured in cm) as the change from baseline (Period 1) over 20 weeks comparing 2 doses of ACM-001.1 with placebo.
  In Arm 3: An evaluation of changes in hip:waist ratio (each circumference measured in cm) as the change from baseline at the end of semaglutide therapy comparing 2 doses of ACM-001.1 with placebo.
Change in body composition (bone mineral composition) during and following semaglutide treatment | 20 weeks
  In Arms 1 & 2: An evaluation of changes in body composition (bone mineral composition (grams/4 weeks)) as the change from baseline (Period 1) over 20 weeks comparing 2 doses of ACM-001.1 with placebo.
  In Arm 3: An evaluation of changes in body composition (bone mineral composition (grams/4 weeks)) as the change from baseline at the end of semaglutide therapy comparing 2 doses of ACM-001.1 with placebo.
Change in body composition (regional lean body mass) during and following semaglutide treatment | 20 Weeks
  In Arms 1 & 2: An evaluation of changes in body composition (regional lean body mass (expressed as grams/4 weeks)) as the change from baseline (Period 1) over 20 weeks comparing 2 doses of ACM-001.1 with placebo.
  In Arm 3: An evaluation of changes in body composition (total and regional lean body mass (expressed as grams/4 weeks)) as the change from baseline at the end of semaglutide therapy comparing 2 doses of ACM-001.1 with placebo.
Evaluation of functional capacity (muscle strength) by stair climbing power (SCP) | 20 weeks
  In Arms 1 & 2: An evaluation of changes in functional capacity (muscle strength) by SCP (SCP/kg) as the change from baseline (Period 1) over 20 weeks comparing 2 doses of ACM-001.1 with placebo.
  In Arm 3: An evaluation of changes in functional capacity (muscle strength) by SCP (SCP/kg) as the change from baseline at the end of semaglutide therapy comparing 2 doses of ACM-001.1 with placebo.
Evaluation of functional capacity (muscle strength) by six minute walk test (6MWT) | 20 Weeks
  In Arms 1 & 2: An evaluation of changes in functional capacity (muscle strength) 6MWT (meters/6 minutes) as the change from baseline (Period 1) over 20 weeks comparing 2 doses of ACM-001.1 with placebo.
  In Arm 3: An evaluation of changes in functional capacity (muscle strength) 6MWT (meters/6 minutes) as the change from baseline at the end of semaglutide therapy comparing 2 doses of ACM-001.1 with placebo.
An evaluation of heart rate (beats/minute) during and following semaglutide treatment | 20 weeks
  In Arms 1 & 2: Heart rate in beats/minute as the change from baseline (Period 1) over 20 weeks comparing 2 doses of ACM-001.1 with placebo.
  In Arm 3: Heart rate in beats/minute as the change from baseline at the end of semaglutide therapy comparing 2 doses of ACM-001.1 with placebo.
An evaluation of electrocardiogram (ECG) abnormalities as change from baseline during and following semaglutide treatment | 20 Weeks
  In Arms 1 & 2: A 12-lead electrocardiogram (ECG) will be performed. The ECG will be reviewed by the Investigator or a qualified designee for abnormalities as change from baseline (Period 1) over 20 weeks comparing 2 doses of ACM-001.1 with placebo. Any medically significant changes from the baseline ECG will be recorded as an AE.
  In Arm 3: A 12-lead ECG will be performed. The ECG will be reviewed by the Investigator or a qualified designee for abnormalities as change from baseline at the end of semaglutide therapy comparing 2 doses of ACM-001.1 with placebo. Any medically significant changes from the baseline ECG will be recorded as an AE.
An evaluation of echocardiogram abnormalities as change from baseline during and following semaglutide treatment | 20 Weeks
  In Arms 1 & 2: An echocardiogram will be performed during the study. The results will be reviewed for abnormalities as change from baseline (Period 1) over 20 weeks comparing 2 doses of ACM-001.1 with placebo. The Investigator responsible for performing the echocardiogram will review the data. Any medically significant changes from the baseline will be recorded as an AE.
  In Arm 3: An echocardiogram will be performed during the study. The results will be reviewed for abnormalities as change from baseline at the end of semaglutide therapy comparing 2 doses of ACM-001.1 with placebo. Any medically significant changes from the baseline will be recorded as an AE.
  On assessment the following data will be collected: left ventricular ejection fraction (LVEF), left ventricular global longitudinal strain (GS), left ventricular end-diastolic diameter (LVEDD), left atrial diameter (LAD) and absolute left ventricular mass (LV mass).
Evaluation of patient reported outcomes during and following semaglutide treatment (quality of life) | 20 weeks
  In Arms 1 & 2: An evaluation of patient reported quality of life assessment by questionnaire as change from baseline (Period 1) over 20 weeks comparing 2 doses of ACM-001.1 with placebo.
  In Arm 3: An evaluation of patient reported quality of life assessment by questionnaire as change from baseline at the end of semaglutide therapy comparing 2 doses of ACM-001.1 with placebo.
Evaluation of patient reported outcomes during and following semaglutide treatment (patient well being) | 20 Weeks
  In Arms 1 & 2: An evaluation of patient reported global assessment of subjective well-being by questionnaire as change from baseline (Period 1) over 20 weeks comparing 2 doses of ACM-001.1 with placebo.
  In Arm 3: An evaluation of patient reported global assessment of subjective well-being by questionnaire as change from baseline at the end of semaglutide therapy comparing 2 doses of ACM-001.1 with placebo.
Evaluation of patient reported outcomes during and following semaglutide treatment (appetite) | 20 Weeks
  In Arms 1 & 2: An evaluation of patient reported appetite using a visual analogue appetite scale as change from baseline (Period 1) over 20 weeks comparing 2 doses of ACM-001.1 with placebo.
  In Arm 3: An evaluation of patient reported appetite using a visual analogue appetite scale as change from baseline at the end of semaglutide therapy comparing 2 doses of ACM-001.1 with placebo.

CONTACTS AND LOCATIONS:
Locations (8):
- Serbia (8):
  - Clinical Hospital Center 'Dr Dragisa Misovic - Dedinje', Belgrade
  - Clinical Hospital Center Bezanijska kosa, Belgrade
  - University Clinical Center of Serbia, Belgrade
  - University Clinical Center Kragujevac, Kragujevac
  - Klinika Za Endocrinologiju, Dijabetes I Bolesti Metabolizma, Niš
  - University Clinical Center of Vojvodina, Novi Sad
  - Opsta bolnica Pancevo, Pančevo
  - Opsta bolnica Valjevo, Valjevo

IPD SHARING:
Plan to Share IPD: Undecided